CLINICAL TRIAL: NCT03203083
Title: Single Leg Squat Performance in Physically and Non-physically Active Individuals: a Cross-sectional Study
Brief Title: Single Leg Squat Performance in Physically and Non-physically Active Individuals
Status: Completed | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: Core Stability L3017
Record Dates: First submitted 2017-06-21; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Single Leg Squat Performance; Athletic Injuries
Keywords: Reproducibility of Results; Clinical Assessment
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- physically active individuals: subjects who perform sports activities more than 6 hours per week
  Interventions: Other: performance of the single leg squat task
- non-physically active individuals: subjects who perform less than 2 hours per week of sport activities
  Interventions: Other: performance of the single leg squat task

INTERVENTIONS:
Other: performance of the single leg squat task — The single-leg squat (SLS) is a clinical functional test commonly used to evaluate clinical abnormal movement patterns of the lower limbs in terms of kinetic chain or co-ordinating muscle activity. This scale accounts for the assessment of five dimensions: overall impression, trunk posture, pelvis in space, hip joint motion and knee join motion. The SLS is potentially promising as a functional test since it involves both daily activity and athletic task.
  Other Names: clinical assessment

SUMMARY:
Single-leg squat (SLS) is a functional test visually rated by clinicians for assessing lower limb function as a preventive injury strategy. SLS clinical rating is a qualitative evaluation and it does not count objective outcomes as kinematics data and surface electromyography (sEMG) assessment. Based on the SLS rating, the aims of this study were (i) to determine the clinical rating agreement among six raters and (ii) to assess kinematic and sEMG predictors of good SLS performance in physically and non-physically active individuals.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) between 18.5-25.5,
* age between 18-35 years old,
* written informed consent to participate,

Exclusion Criteria:

- musculoskeletal pain or history of lower extremity injuries lasting more than three months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A cohort of healthy young subjects was recruited.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2014-03-19 (Actual); Primary Completion 2014-07-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
reliability of the clinical assessment | Baseline
  intra- and inter-rater reliability for six clinicians when performing the SLS clinical rating assessment
reliability of the clinical assessment | 2 weeks after the first evaluation
  intra- and inter-rater reliability for six clinicians when performing the SLS clinical rating assessment
reliability of the clinical assessment | 1 month after the first evaluation
  intra- and inter-rater reliability for six clinicians when performing the SLS clinical rating

SECONDARY OUTCOMES:
kinematic predictors | Baseline
  The following kinematic variables were considered during the single-leg squat: ipsilateral hip flexion in the lateral plane, hip internal rotation, hip adduction, pelvic obliquity, knee flexion (lateral plane) and medio-lateral displacement (frontal plane).
sEMG predictors | Baseline
  The surface Electromyography (sEMG) activity of the following muscles were assessed: tensor fasciae latae, rectus femoris, adductor longus, gluteus maximus and transversus abdominis.

REFERENCES:
- [Derived] Gianola S, Castellini G, Stucovitz E, Nardo A, Banfi G. Single leg squat performance in physically and non-physically active individuals: a cross-sectional study. BMC Musculoskelet Disord. 2017 Jul 14;18(1):299. doi: 10.1186/s12891-017-1660-8. PMID 28709418